CLINICAL TRIAL: NCT07174011
Title: Evaluation of the Efficacy and Safety of Oral Roflumilast Versus Intralesional Corticosteroids Injection (ILCs) in the Treatment of Alopecia Areata: A Randomized Controlled Trial.
Brief Title: Evaluation of the Efficacy and Safety of Oral Roflumilast Versus Intralesional Corticosteroids Injection (ILCs) in the Treatment of Alopecia Areata
Acronym: AA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Maher Mahmoud Mahran, Lecturer of Dermatology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-79-2025
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Alopecia; Alopecia Areata
Keywords: Intralesional Corticosteroids Injection (ILCs); Roflumilast; Alopecia areata
MeSH Terms: conditions — Alopecia; Alopecia Areata | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: 25 participants with AA will be on Roflumilast group (Active Comparator): patients in arm A will receive daily oral Roflumilast (immunomodulator) 500 mcg for 16Consecutive weeks.
  Interventions: Drug: Roflumilast
- 25 participants will receive intralesional steroid injection (Active Comparator): ILCs group: 5 mg/mL every 4 weeks for 16 weeks
  Interventions: Drug: intralesional steroid

INTERVENTIONS:
Drug: Roflumilast — Phosphodiesterase-4 (PDE4) inhibitor assigned to arm A
  Arms: Arm A: 25 participants with AA will be on Roflumilast group
Drug: intralesional steroid — intralesional injection of corticosteroid
  Arms: 25 participants will receive intralesional steroid injection

SUMMARY:
Evaluation of the Efficacy and Safety of a drug called Oral Roflumilast versus Intralesional Corticosteroids Injection (ILCs) in the Treatment of Alopecia Areata.

DETAILED DESCRIPTION:
we are going to evaluate using oral immunomodulator called Roflumilast and compare its safety and efficacy to intralesional steroid injection in the treatment of Alopecia areata

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate patchy alopecia areata as assessed by SALT score (S1: 1-24% hair loss (limited); S2: 25-49% hair loss (moderate))
* Patients with patchy alopecia areata with viable hair follicles by trichoscopy.
* Patients of both genders aged >18 years.
* Patients able and willing to provide informed consent.

Exclusion Criteria:

* Patients with other types of AA (surface area >50%, alopecia totalis, alopecia universalis and ophiasis).
* Patients less than 18 years old.
* Patients receiving systemic treatment relevant to AA or biologics, phototherapy, or topical treatment within 4 weeks before enrollment into the study.
* Patients with a history of/ or existing scalp skin diseases apart from AA, such as eczema, seborrheic dermatitis, psoriasis, scalp infections, or skin cancer.
* Pregnant and lactating females.
* Patients with a history of other inflammatory skin conditions
* History of hypersensitivity to roflumilast or its components.
* History of severe anxiety or depression (Gupta, 2012)
* Patients with history of bleeding disorders or on anticoagulant medications,
* Patients with active infection at the local site, patients with keloidal tendency, and patients with low pain threshold.

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
To assess the degree of improvement in hair regrowth according to the change in SALT score from baseline to Week 16. | 4 months
  To assess the degree of improvement in hair regrowth according to the change in SALT score from baseline to Week 16.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
age, sex